CLINICAL TRIAL: NCT01410149
Title: The Influence of Mode and Patient-ventilator Interaction on Sleep Quality in the ICU
Brief Title: Sleep Quality in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Lung Association (Other); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Karen Bosma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R-07-106; 13114 (Other: REB)
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Respiratory Failure
Keywords: PAV (proportional assist ventilation); sleep; polysomnography; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PAV (Active Comparator): Proportional Assist Ventilation (PAV+ on PB840 ventilator)
  Interventions: Other: PAV
- PSV (Active Comparator): Pressure Support Ventilation (PSV on PB840 ventilator)
  Interventions: Other: PSV
- ACV (Active Comparator): Assist Control/ Pressure limited Ventilation (on PB840 ventilator)
  Interventions: Other: ACV

INTERVENTIONS:
Other: PAV — Proportional Assist Ventilation will be used to ventilate the patient for a 24 hour period
  Arms: PAV
Other: PSV — Pressure Support Ventilation will be used to ventilate the patient for a 24 hour period
  Arms: PSV
Other: ACV — Assist Control Ventilation will be used to ventilate the patient for a 24 hour period
  Arms: ACV

SUMMARY:
Patients requiring mechanical ventilation in the ICU will undergo three consecutive nights of polysomnography to record sleep patterns while receiving three modes of mechanical ventilation; Proportional assist ventilation (PAV), Pressure support ventilation (PSV), Assist control ventilation (ACV), applied in random order. The purpose is to determine the effect of mode of mechanical ventilation on patient-ventilator asynchrony and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* received mechanical ventilation >72 hours
* glasgow coma scale >10
* acute physiology score <13
* ready for partial ventilatory support: intact respiratory drive, PaO2/FiO2 ratio >200 on positive end expiratory pressure (PEEP) less than or equal to 5 cmH2O, and PH of 7.35 to 7.45
* sedation: analgesia at dose not higher than 0.01 mg/kg/hr morphine equivalent x 48 hours, sedation at dose not higher than 0.01 mg/kg/hr lorazepam equivalent x 72 hours.
* anticipate ongoing need for partial ventilatory support for the following 72 hours

Exclusion Criteria:

* Successful completion of spontaneous breathing trial
* Neurological injury, encephalopathy or abnormal EEG
* History of central sleep apnea
* General anaesthesia within 72 hours from study entry
* Requiring haloperidol >10 mg/24 hours
* hemodynamically unstable
* sepsis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 3 nights
  Sleep fragmentation (number of arousals and awakenings/hr sleep), sleep architecture (% time asleep spent in Stage 1, 2, 3/4 and REM sleep)

SECONDARY OUTCOMES:
Patient-ventilator asynchrony | 3 nights
  Incidence of patient-ventilator asynchrony (asynchrony index, % of asynchronous breaths per minute)

OTHER OUTCOMES:
Delirium | 3 days
  Positive score on a delirium screening tool (CAM-ICU or ICDSC)
Comfort | 3 days
  Patient's assessment of their own breathing comfort and their perceived quality of sleep, indicated on a visual analogue scale
Respiratory pattern | 3 nights
  Measurement of average tidal volume, respiratory rate, minute ventilation and non-invasive measurement of respiratory muscle effort relative to maximum effort
Blood gas | evening and morning
  measurement of paO2 and paCO2

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Bosma, MD, FRCPC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Parthasarathy S. Effects of sleep on patient-ventilator interaction. Respir Care Clin N Am. 2005 Jun;11(2):295-305. doi: 10.1016/j.rcc.2005.02.004. PMID 15936695
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Parthasarathy S. Sleep during mechanical ventilation. Curr Opin Pulm Med. 2004 Nov;10(6):489-94. doi: 10.1097/01.mcp.0000143691.94442.fa. PMID 15510055
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Irwin M, McClintick J, Costlow C, Fortner M, White J, Gillin JC. Partial night sleep deprivation reduces natural killer and cellular immune responses in humans. FASEB J. 1996 Apr;10(5):643-53. doi: 10.1096/fasebj.10.5.8621064.
- [Background] Chen HI, Tang YR. Sleep loss impairs inspiratory muscle endurance. Am Rev Respir Dis. 1989 Oct;140(4):907-9. doi: 10.1164/ajrccm/140.4.907. PMID 2802378
- [Background] Helton MC, Gordon SH, Nunnery SL. The correlation between sleep deprivation and the intensive care unit syndrome. Heart Lung. 1980 May-Jun;9(3):464-8. No abstract available. PMID 6901518
- [Background] Parthasarathy S, Tobin MJ. Effect of ventilator mode on sleep quality in critically ill patients. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1423-9. doi: 10.1164/rccm.200209-999OC. Epub 2002 Sep 5. PMID 12406837
- [Background] Fanfulla F, Delmastro M, Berardinelli A, Lupo ND, Nava S. Effects of different ventilator settings on sleep and inspiratory effort in patients with neuromuscular disease. Am J Respir Crit Care Med. 2005 Sep 1;172(5):619-24. doi: 10.1164/rccm.200406-694OC. Epub 2005 Jun 16. PMID 15961699
- [Background] Bosma K, Ferreyra G, Ambrogio C, Pasero D, Mirabella L, Braghiroli A, Appendini L, Mascia L, Ranieri VM. Patient-ventilator interaction and sleep in mechanically ventilated patients: pressure support versus proportional assist ventilation. Crit Care Med. 2007 Apr;35(4):1048-54. doi: 10.1097/01.CCM.0000260055.64235.7C. PMID 17334259
- [Background] Meza S, Mendez M, Ostrowski M, Younes M. Susceptibility to periodic breathing with assisted ventilation during sleep in normal subjects. J Appl Physiol (1985). 1998 Nov;85(5):1929-40. doi: 10.1152/jappl.1998.85.5.1929. PMID 9804601
- [Background] Younes M. Proportional assist ventilation, a new approach to ventilatory support. Theory. Am Rev Respir Dis. 1992 Jan;145(1):114-20. doi: 10.1164/ajrccm/145.1.114. PMID 1731573